CLINICAL TRIAL: NCT04236479
Title: Mesenchymal Stromal Cells Delivery Through Cardiopulmonary Bypass in Pediatric Cardiac Surgery
Brief Title: Mesenchymal Stromal Cells for Infants With Congenital Heart Disease (MedCaP)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director, Center for Cancer and Immunology/ Center for Emerging Technologies in Immune Cell Therapies (CETI), Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011914
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease (CHD)
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone marrow-derived mesenchymal stromal cell (BM-MSC) (Experimental): The dose-escalation methods with a modified continual reassessment at the five dose levels (1x10^6, 10x10^6, 20x10^6, 40x10^6, 80x10^6 cells/kg) will be performed to determine safety and feasibility of allogeneic BM-MSC infusion during pediatric cardiac surgery and the maximum tolerated dose in infants with CHD.
  Interventions: Biological: BM-MSC

INTERVENTIONS:
Biological: BM-MSC — Allogeneic bone marrow-derived mesenchymal stromal cell (BM-MSC) delivery through cardiopulmonary bypass (CPB) using a homogeneous population of infants with congenital heart disease (CHD) who will be undergoing a two-ventricle repair within the first six months of life.

SUMMARY:
The proposed study will be a prospective, open-label, single-center, safety and feasibility phase 1 trial of allogeneic bone marrow-derived mesenchymal stromal cell (BM-MSC) delivery though cardiopulmonary bypass (CPB) using a homogeneous population of infants with congenital heart disease (CHD) who will be undergoing a two-ventricle repair within the first six months of life

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-center, safety and feasibility phase 1 trial of allogeneic bone marrow-derived mesenchymal stromal cell (BM-MSC) delivery though cardiopulmonary bypass (CPB) using a homogeneous population of infants with congenital heart disease (CHD) who will be undergoing a two-ventricle repair within the first six months of life. The dose-escalation methods with a modified continual reassessment at the five dose levels (1x10^6, 10x10^6, 20x10^6, 40x10^6, 80x10^6, cells/kg) will be performed to determine safety and feasibility of allogeneic BM-MSC infusion during pediatric cardiac surgery and the maximum tolerated dose in infants with CHD. In addition to the primary objective of assessing the safety and feasibility of BM-MSC delivery through CPB, our secondary objectives are designed to develop biological signature measures and clinical outcome measures feasible for use in larger efficacy and effectiveness trials with a particular focus on neurodevelopmental outcome and early postoperative course after BM-MSC treatment. We will determine actual magnitude of differences in neuroimaging and neurodevelopmental variables and postoperative inflammatory and pathophysiological variables after BM-MSC delivery in infants with CHD. Enrollment, follow-up, and analysis are planned to occur over 36 months for the treatment and initial follow-up portions of the study. Long-term follow-up until 18 months of age will be subsequently reported.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal and young infantile patients who are ≤ 3 months of age
* Scheduled to undergo reparative two-ventricle repair for congenital heart defects without aortic arch reconstruction, including the following:

  a. D-Transposition of the Great Arteries (d-TGA) Group: i. d-TGA with intact ventricular septum (d-TGA, IVS) ii. d-TGA with ventricular septal defect (d-TGA, VSD) b. Ventricular Septal Defect (VSD) Group: i. VSD without aortic arch obstruction (AAO) ii. Complete common atrioventricular canal defect (CAVC) c. Tetralogy of Fallot (TOF) Group: i. Tetralogy of Fallot (TOF) ii. Tetralogy of Fallot with Pulmonary Atresia (TOF,PA) iii. Truncus arteriosus (TA) iv. Double outlet right ventricle (DORV)
* Scheduled surgery at or before three months of age.
* Parent/guardian capable of providing informed consent.

Exclusion Criteria:

* Birth weight less than 2.0 kg
* Recognizable phenotypic syndrome
* Associated extracardiac anomalies of greater than minor severity
* Previous cardiac surgery
* Associated cardiovascular anomalies requiring aortic arch reconstruction and/or additional open cardiac surgical procedures in infancy
* Prior severe hypoxic event
* Significant screening test values that place subjects at increased risk of complications from participation in the study

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who experience serious adverse events, adverse events, and/or early treatment discontinuations. | 45 days following the MSC administration
  Dose Limiting Toxicity is attributable to the MSC administration.

SECONDARY OUTCOMES:
Actual magnitude of differences in neuroimaging and neurodevelopmental variables will be measured after MSC delivery. | 18 months
  Secondary objective will be measured by using the Pediatric Cardiac Critical Care Consortium (PC4) registry system.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jonas, MD, Principal Investigator — CNMC
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No